CLINICAL TRIAL: NCT06562439
Title: Early Identification and Intervention Of Developmental Delay Among Infants And Toddlers With Sickle Cell Disease Using the Sickle Cell Caregiver Collaboration for Child Development (SCCCD) Intervention
Brief Title: Testing the Sickle Cell Caregiver Collaboration for Child Development (SCCCD) Intervention
Acronym: SCCCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCCCD.SRP.OT; K23HL161328 (NIH)
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease
Keywords: child development; developmental delay; parents as teachers; home based intervention
MeSH Terms: conditions — Anemia, Sickle Cell; Learning Disabilities | interventions — Child Development

STUDY DESIGN:
Intervention Model Description: We will randomize children to receive developmental screening alone or developmental screening with a home-based intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developmental Screening (No Intervention): Participants in this group will complete developmental screening at 9, 18, and 30 months of age.
- Developmental Screening + Home-Based Intervention (Experimental): Participants in this group will complete developmental screening at 9, 18 and 30 months of age and monthly home visits with the family using the Parents as Teachers curriculum.
  Interventions: Behavioral: Sickle Cell Collaboration for Child Development

INTERVENTIONS:
Behavioral: Sickle Cell Collaboration for Child Development — The Sickle Cell Collaboration for Child Development (SCCCD) combines the Parents as Teachers curriculum with experienced occupational therapy to help families and children meet their learning and developmental goals.
  Arms: Developmental Screening + Home-Based Intervention

SUMMARY:
Sickle cell disease affects 100,000 people and 2,000 newborns each year; 50% of these children have a developmental deficit (>2 SD) before the age of 3. Early identification of developmental deficit supports timely intervention, but children with sickle cell disease are grossly underdiagnosed and undertreated. The goal of the proposed study is to determine the incidence and severity of developmental deficit at 9, 18 and 30 months of age among children with sickle cell disease and test a 12-month, home-based caregiver intervention with this disproportionately affected population.

DETAILED DESCRIPTION:
This trial will be conducted in two phases. In Aim 1, the investigators are evaluating the developmental progress of children with and without sickle cell disease (SCD) at 9, 18, and 30 months. The investigators aim to recruit a total of 100 children and their caregivers (SCD = 50, Comparison = 50). Each child/caregiver dyad will be asked to complete 3 evaluation visits where the child's developmental progress will be evaluated and the caregiver will complete surveys related to their child's development, participation, and the caregiver's mental health.

In Aim 2, children with sickle cell disease will be randomized to receive developmental evaluations at 9, 18, and 30 months alone or a 12-month home-based intervention + developmental evaluations. The intervention is called the Sickle Cell Collaboration for Child Development (SCCCD) uses the widely used Parents as Teachers curriculum and is supplemented with specific support for the caregivers related to the child's sickle cell diagnosis. This pilot randomized controlled trial design is designed to (1) examine the potential effects of SCCCD on child development and caregiver well-being compared to the group with no intervention and (2) optimize trial procedures to enhance acceptability and scalability in preparation for a full-scale trial. Data will be collected to explore determinants (facilitators and barriers) affecting participation and outcomes. The investigators will recruit 50 children with sickle cell disease to this aim, with the goal to have 25 children randomized to intervention. Randomization will be completed using a random computer generator that can balance groups based on key factors like age, sex, and area deprivation index (index approximating income and community resources).

Participants randomized to SCCCD (n=25) will be invited to participate in 12 home-based intervention session over the course of 1 year (1 visit monthly) with a trained parent educator. They will complete the visit according to the Parents as Teachers curriculum and will provide additional discussion focused on sickle cell disease and strategies to promote child development. If caregivers are uncomfortable with home-visits, families will have the option to complete intervention visits in our on-site clinic space or in a preferred community location (e.g., public library, child care setting, place of worship). Participants in the developmental evaluation group will complete study visits as described in Aim 1.

The primary outcomes are child development and caregiver acceptability of developmental screening and intervention. The investigators will use implementation strategies guided by our earlier work to optimize the program's feasibility which will be measured by tracking participation and retention rates in each phase of this study. Acceptability will be assessed through interviews and surveys.

ELIGIBILITY:
Inclusion Criteria:

* All sickle cell disease genotypes will be included. Children will be eligible to participate until they reach 31 months of age (1 month over target evaluation).

Exclusion Criteria:

* Children will be excluded if the child has fragile health, a diagnosis associated with developmental deficit (not sickle cell disease), or the family is not English language proficient -because of limitations in alternative language assessment and intervention delivery.

Ages: 6 Months to 31 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant Toddler Development-IV | Completed at 9, 18 and 30 months
  Child participants will complete up to 3 developmental evaluations with a trained evaluator using the Bayley Scales of Infant Toddler Development-IV. The Bayley assesses development in the domains of cognition, fine and gross motor, and expressive and receptive language. Caregiver questionnaires assess adaptive behavior and social emotional development. Scaled scores range from 1-19, where a score of 10 is average and a higher score indicates better outcome.
Ages and Stages Questionnaire-3 | Completed at 9, 18 and 30 months
  Caregivers will complete the Ages and Stages Questionnaire-3, which assesses the caregivers perspective of how their child is meeting developmental milestones in the domains of communication, gross motor, fine motor, personal-social and problem solving. Scores range from 0-60, where a higher score indicates a better outcome.
Infant Toddler Activity Card Sort | Completed at 9, 18 and 30 months
  Caregivers will complete the Infant Toddler Activity Card Sort (ITACS) to determine activities and routines that are presenting performance or participation challenges for families in the context of their everyday lives.
Behavior Rating Inventory of Executive Function-Preschool | 30 months of age
  The Behavior Rating Inventory of Executive Function-Preschool (BRIEF) evaluates executive functioning of toddlers >2.5 years. Executive functioning is identified as a high risk domain for deficits among individuals with sickle cell disease. Raw scores are converted to t-scores (mean = 50, SD = 10) and scores above 65 are considered clinically significant.

SECONDARY OUTCOMES:
PROMIS Depression (Caregiver) | Completed at child's 9, 18 and 30 month evaluation.
  The Patient Reported Outcomes Measurement Information Systems (PROMIS) Depression short form is a valid and reliable 8-item tool to screen for depression. Scores range from 8-40, with higher scores indicating more severe depression symptoms.
Acceptability | through study completion, an average of 1 year
  Study visit completion rates and notes from intervention visits will be reviewed. Interviews will be conducted with all participants in the SCCCD intervention, regardless of completion to determine components that contributed to participation or attrition.
Fidelity | through study completion, an average of 1 year
  The Comprehensive Intervention Fidelity Guide will be used to evaluate intervention design, training and delivery. This guide specifies the intervention model, the fidelity indices (e.g., participation and retention rates) and compare those to outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Findings from this proposal will be disseminated in peer-reviewed publications and at scholarly meetings following best practices guidelines (e.g., Equator network guidelines).

REFERENCES:
- [Background] Brownson RC, Proctor EK, Luke DA, Baumann AA, Staub M, Brown MT, Johnson M. Building capacity for dissemination and implementation research: one university's experience. Implement Sci. 2017 Aug 16;12(1):104. doi: 10.1186/s13012-017-0634-4. PMID 28814328
- [Background] Campbell FA, Ramey CT. Effects of early intervention on intellectual and academic achievement: a follow-up study of children from low-income families. Child Dev. 1994 Apr;65(2 Spec No):684-98. PMID 8013248
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Hennink M, Kaiser BN. Sample sizes for saturation in qualitative research: A systematic review of empirical tests. Soc Sci Med. 2022 Jan;292:114523. doi: 10.1016/j.socscimed.2021.114523. Epub 2021 Nov 2. PMID 34785096
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Nilsen P, Bernhardsson S. Context matters in implementation science: a scoping review of determinant frameworks that describe contextual determinants for implementation outcomes. BMC Health Serv Res. 2019 Mar 25;19(1):189. doi: 10.1186/s12913-019-4015-3. PMID 30909897
- [Background] Toomey E, Hardeman W, Hankonen N, Byrne M, McSharry J, Matvienko-Sikar K, Lorencatto F. Focusing on fidelity: narrative review and recommendations for improving intervention fidelity within trials of health behaviour change interventions. Health Psychol Behav Med. 2020 Mar 12;8(1):132-151. doi: 10.1080/21642850.2020.1738935. PMID 34040865
- [Background] Nelson MC, Cordray DS, Hulleman CS, Darrow CL, Sommer EC. A procedure for assessing intervention fidelity in experiments testing educational and behavioral interventions. J Behav Health Serv Res. 2012 Oct;39(4):374-96. doi: 10.1007/s11414-012-9295-x. PMID 22935907
- [Background] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Background] Pilkonis PA, Yu L, Dodds NE, Johnston KL, Maihoefer CC, Lawrence SM. Validation of the depression item bank from the Patient-Reported Outcomes Measurement Information System (PROMIS) in a three-month observational study. J Psychiatr Res. 2014 Sep;56:112-9. doi: 10.1016/j.jpsychires.2014.05.010. Epub 2014 May 29. PMID 24931848
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Hoyt CR, L'Hotta AJ, Bauer AH, Chang CH, Varughese TE, Abel RA, King AA. Activity competence among infants and toddlers with developmental disabilities: Rasch analysis of the Infant Toddler Activity Card Sort (ITACS). J Patient Rep Outcomes. 2021 Jan 21;5(1):14. doi: 10.1186/s41687-021-00287-0. PMID 33475869
- [Background] Schatz J, Roberts CW. Neurobehavioral impact of sickle cell disease in early childhood. J Int Neuropsychol Soc. 2007 Nov;13(6):933-43. doi: 10.1017/S1355617707071196. PMID 17942011
- [Background] Rydz D, Srour M, Oskoui M, Marget N, Shiller M, Birnbaum R, Majnemer A, Shevell MI. Screening for developmental delay in the setting of a community pediatric clinic: a prospective assessment of parent-report questionnaires. Pediatrics. 2006 Oct;118(4):e1178-86. doi: 10.1542/peds.2006-0466. PMID 17015506
- [Background] Radecki L, Sand-Loud N, O'Connor KG, Sharp S, Olson LM. Trends in the use of standardized tools for developmental screening in early childhood: 2002-2009. Pediatrics. 2011 Jul;128(1):14-9. doi: 10.1542/peds.2010-2180. Epub 2011 Jun 27. PMID 21708798
- [Background] Hoyt CR, Chuck AC, Varughese TE, Fisher LC, Manis HE, O'Connor KE, Shen E, Wong AWK, Abel RA, King AA. Psychometric Properties of the Infant Toddler Activity Card Sort. OTJR (Thorofare N J). 2021 Oct;41(4):259-267. doi: 10.1177/15394492211012657. Epub 2021 May 6. PMID 33955289
- [Background] Hoyt CR, Fernandez JD, Varughese TE, Grandgeorge E, Manis HE, O'Connor KE, Abel RA, King AA. The Infant Toddler Activity Card Sort: A Caregiver Report Measure of Children's Occupational Engagement in Family Activities and Routines. OTJR (Thorofare N J). 2020 Jan;40(1):36-41. doi: 10.1177/1539449219852030. Epub 2019 Jun 4. PMID 31161868
- [Background] Kind AJH, Buckingham WR. Making Neighborhood-Disadvantage Metrics Accessible - The Neighborhood Atlas. N Engl J Med. 2018 Jun 28;378(26):2456-2458. doi: 10.1056/NEJMp1802313. No abstract available. PMID 29949490
- [Background] Heitzer AM, Cohen DL, Okhomina VI, Trpchevska A, Potter B, Longoria J, Porter JS, Estepp JH, King A, Henley M, Kang G, Hankins JS. Neurocognitive functioning in preschool children with sickle cell disease. Pediatr Blood Cancer. 2022 Mar;69(3):e29531. doi: 10.1002/pbc.29531. Epub 2021 Dec 31. PMID 34971013
- [Background] Hogan AM, Pit-ten Cate IM, Vargha-Khadem F, Prengler M, Kirkham FJ. Physiological correlates of intellectual function in children with sickle cell disease: hypoxaemia, hyperaemia and brain infarction. Dev Sci. 2006 Jul;9(4):379-87. doi: 10.1111/j.1467-7687.2006.00503.x. PMID 16764611
- [Background] Olds DL, Robinson J, O'Brien R, Luckey DW, Pettitt LM, Henderson CR Jr, Ng RK, Sheff KL, Korfmacher J, Hiatt S, Talmi A. Home visiting by paraprofessionals and by nurses: a randomized, controlled trial. Pediatrics. 2002 Sep;110(3):486-96. doi: 10.1542/peds.110.3.486. PMID 12205249
- [Background] Olds DL, Sadler L, Kitzman H. Programs for parents of infants and toddlers: recent evidence from randomized trials. J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):355-91. doi: 10.1111/j.1469-7610.2006.01702.x. PMID 17355402
- [Background] Wagner MM, Clayton SL. The Parents as Teachers program: results from two demonstrations. Future Child. 1999 Spring-Summer;9(1):91-115, 179-89. PMID 10414012
- [Background] Bann CM, Wallander JL, Do B, Thorsten V, Pasha O, Biasini FJ, Bellad R, Goudar S, Chomba E, McClure E, Carlo WA. Home-Based Early Intervention and the Influence of Family Resources on Cognitive Development. Pediatrics. 2016 Apr;137(4):e20153766. doi: 10.1542/peds.2015-3766. Epub 2016 Mar 14. PMID 26977079
- [Background] Neuhauser A, Ramseier E, Schaub S, Burkhardt SCA, Lanfranchi A. MEDIATING ROLE OF MATERNAL SENSITIVITY: ENHANCING LANGUAGE DEVELOPMENT IN AT-RISK FAMILIES. Infant Ment Health J. 2018 Sep;39(5):522-536. doi: 10.1002/imhj.21738. Epub 2018 Aug 8. PMID 30088285
- [Background] Chaiyachati BH, Gaither JR, Hughes M, Foley-Schain K, Leventhal JM. Preventing child maltreatment: Examination of an established statewide home-visiting program. Child Abuse Negl. 2018 May;79:476-484. doi: 10.1016/j.chiabu.2018.02.019. Epub 2018 Mar 20. PMID 29558714
- [Background] Yarboi J, Prussien KV, Bemis H, Williams E, Watson KH, McNally C, Henry L, King AA, DeBaun MR, Compas BE. Responsive Parenting Behaviors and Cognitive Function in Children With Sickle Cell Disease. J Pediatr Psychol. 2019 Nov 1;44(10):1234-1243. doi: 10.1093/jpepsy/jsz065. PMID 31579920
- [Background] Thompson RJ Jr, Gustafson KE, Bonner MJ, Ware RE. Neurocognitive development of young children with sickle cell disease through three years of age. J Pediatr Psychol. 2002 Apr-May;27(3):235-44. doi: 10.1093/jpepsy/27.3.235. PMID 11909931
- [Background] Varughese TE, Hoyt CR, L'Hotta AJ, Ikemenogo PA, Howdeshell SG, Housten AJ, Abel RA, King AA. Stress and the Home Environment in Caregivers of Children with Sickle Cell. J Pediatr Psychol. 2020 Jun 1;45(5):521-529. doi: 10.1093/jpepsy/jsaa016. PMID 32232470
- [Background] Committee on Children With Disabilities. Role of the pediatrician in family-centered early intervention services. Pediatrics. 2001 May;107(5):1155-7. doi: 10.1542/peds.107.5.1155. PMID 11331701
- [Background] Gallegos A, Dudovitz R, Biely C, Chung PJ, Coker TR, Barnert E, Guerrero AD, Szilagyi PG, Nelson BB. Racial Disparities in Developmental Delay Diagnosis and Services Received in Early Childhood. Acad Pediatr. 2021 Sep-Oct;21(7):1230-1238. doi: 10.1016/j.acap.2021.05.008. Epub 2021 May 19. PMID 34020100
- [Background] Shook LM, Farrell CB, Kalinyak KA, Nelson SC, Hardesty BM, Rampersad AG, Saving KL, Whitten-Shurney WJ, Panepinto JA, Ware RE, Crosby LE. Translating sickle cell guidelines into practice for primary care providers with Project ECHO. Med Educ Online. 2016 Nov 24;21:33616. doi: 10.3402/meo.v21.33616. eCollection 2016. PMID 27887664
- [Background] Whiteman LN, Haywood C Jr, Lanzkron S, Strouse JJ, Feldman L, Stewart RW. Primary Care Providers' Comfort Levels in Caring for Patients with Sickle Cell Disease. South Med J. 2015 Sep;108(9):531-6. doi: 10.14423/SMJ.0000000000000331. PMID 26332477
- [Background] Lipkin PH, Macias MM, Baer Chen B, Coury D, Gottschlich EA, Hyman SL, Sisk B, Wolfe A, Levy SE. Trends in Pediatricians' Developmental Screening: 2002-2016. Pediatrics. 2020 Apr;145(4):e20190851. doi: 10.1542/peds.2019-0851. Epub 2020 Mar 2. PMID 32123018
- [Background] Armstrong FD, Elkin TD, Brown RC, Glass P, Rana S, Casella JF, Kalpatthi RV, Pavlakis S, Mi Z, Wang WC; Baby Hug Investigators. Developmental function in toddlers with sickle cell anemia. Pediatrics. 2013 Feb;131(2):e406-14. doi: 10.1542/peds.2012-0283. Epub 2013 Jan 6. PMID 23296434
- [Background] Drazen CH, Abel R, Gabir M, Farmer G, King AA. Prevalence of Developmental Delay and Contributing Factors Among Children With Sickle Cell Disease. Pediatr Blood Cancer. 2016 Mar;63(3):504-10. doi: 10.1002/pbc.25838. Epub 2015 Nov 17. PMID 26575319
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Wang WC, Zou P, Hwang SN, Kang G, Ding J, Heitzer AM, Schreiber JE, Helton K, Hankins JS. Effects of hydroxyurea on brain function in children with sickle cell anemia. Pediatr Blood Cancer. 2021 Oct;68(10):e29254. doi: 10.1002/pbc.29254. Epub 2021 Jul 31. PMID 34331507
- [Background] Miller M, Landsman R, Scott JP, Heffelfinger AK. Fostering equity in education and academic outcomes in children with sickle cell disease. Clin Neuropsychol. 2022 Feb;36(2):245-263. doi: 10.1080/13854046.2021.1945147. Epub 2021 Jul 5. PMID 34218732
- [Background] Burnes DP, Antle BJ, Williams CC, Cook L. Mothers raising children with sickle cell disease at the intersection of race, gender, and illness stigma. Health Soc Work. 2008 Aug;33(3):211-20. doi: 10.1093/hsw/33.3.211. PMID 18773796
- [Background] Nelson SC, Hackman HW. Race matters: perceptions of race and racism in a sickle cell center. Pediatr Blood Cancer. 2013 Mar;60(3):451-4. doi: 10.1002/pbc.24361. Epub 2012 Sep 28. PMID 23023789
- [Background] Constantino JN, Abbacchi AM, Saulnier C, Klaiman C, Mandell DS, Zhang Y, Hawks Z, Bates J, Klin A, Shattuck P, Molholm S, Fitzgerald R, Roux A, Lowe JK, Geschwind DH. Timing of the Diagnosis of Autism in African American Children. Pediatrics. 2020 Sep;146(3):e20193629. doi: 10.1542/peds.2019-3629. PMID 32839243
- [Background] Schatz J, Schlenz AM, Smith KE, Roberts CW. Predictive validity of developmental screening in young children with sickle cell disease: a longitudinal follow-up study. Dev Med Child Neurol. 2018 May;60(5):520-526. doi: 10.1111/dmcn.13689. Epub 2018 Feb 28. PMID 29488622
- [Background] Schatz J, McClellan CB, Puffer ES, Johnson K, Roberts CW. Neurodevelopmental screening in toddlers and early preschoolers with sickle cell disease. J Child Neurol. 2008 Jan;23(1):44-50. doi: 10.1177/0883073807307982. Epub 2007 Dec 26. PMID 18160556
- [Background] Hogan AM, Kirkham FJ, Prengler M, Telfer P, Lane R, Vargha-Khadem F, Haan M. An exploratory study of physiological correlates of neurodevelopmental delay in infants with sickle cell anaemia. Br J Haematol. 2006 Jan;132(1):99-107. doi: 10.1111/j.1365-2141.2005.05828.x. PMID 16371025
- [Background] Kawadler JM, Clayden JD, Clark CA, Kirkham FJ. Intelligence quotient in paediatric sickle cell disease: a systematic review and meta-analysis. Dev Med Child Neurol. 2016 Jul;58(7):672-9. doi: 10.1111/dmcn.13113. Epub 2016 Mar 31. PMID 27038278
- [Background] Prussien KV, Jordan LC, DeBaun MR, Compas BE. Cognitive Function in Sickle Cell Disease Across Domains, Cerebral Infarct Status, and the Lifespan: A Meta-Analysis. J Pediatr Psychol. 2019 Sep 1;44(8):948-958. doi: 10.1093/jpepsy/jsz031. PMID 31050352
- [Background] Damschroder LJ, Reardon CM, Opra Widerquist MA, Lowery J. Conceptualizing outcomes for use with the Consolidated Framework for Implementation Research (CFIR): the CFIR Outcomes Addendum. Implement Sci. 2022 Jan 22;17(1):7. doi: 10.1186/s13012-021-01181-5. PMID 35065675
- [Background] Davis M, Beidas RS. Refining contextual inquiry to maximize generalizability and accelerate the implementation process. Implement Res Pract. 2021 Mar 17;2:2633489521994941. doi: 10.1177/2633489521994941. eCollection 2021 Jan-Dec. PMID 37089986
- [Background] Council on Children With Disabilities; Section on Developmental Behavioral Pediatrics; Bright Futures Steering Committee; Medical Home Initiatives for Children With Special Needs Project Advisory Committee. Identifying infants and young children with developmental disorders in the medical home: an algorithm for developmental surveillance and screening. Pediatrics. 2006 Jul;118(1):405-20. doi: 10.1542/peds.2006-1231. PMID 16818591
- [Background] DeBaun MR, Jordan LC, King AA, Schatz J, Vichinsky E, Fox CK, McKinstry RC, Telfer P, Kraut MA, Daraz L, Kirkham FJ, Murad MH. American Society of Hematology 2020 guidelines for sickle cell disease: prevention, diagnosis, and treatment of cerebrovascular disease in children and adults. Blood Adv. 2020 Apr 28;4(8):1554-1588. doi: 10.1182/bloodadvances.2019001142. PMID 32298430
- [Background] Proctor EK, Powell BJ, McMillen JC. Implementation strategies: recommendations for specifying and reporting. Implement Sci. 2013 Dec 1;8:139. doi: 10.1186/1748-5908-8-139. PMID 24289295
- [Background] Hoyt Drazen C, Abel R, Lindsey T, King AA. Development and feasibility of a home-based education model for families of children with sickle cell disease. BMC Public Health. 2014 Feb 5;14:116. doi: 10.1186/1471-2458-14-116. PMID 24499305
- [Background] Peacock S, Konrad S, Watson E, Nickel D, Muhajarine N. Effectiveness of home visiting programs on child outcomes: a systematic review. BMC Public Health. 2013 Jan 9;13:17. doi: 10.1186/1471-2458-13-17. PMID 23302300
- [Background] King AA, Rodeghier MJ, Panepinto JA, Strouse JJ, Casella JF, Quinn CT, Dowling MM, Sarnaik SA, Thompson AA, Woods GM, Minniti CP, Redding-Lallinger RC, Kirby-Allen M, Kirkham FJ, McKinstry R, Noetzel MJ, White DA, Kwiatkowski JK, Howard TH, Kalinyak KA, Inusa B, Rhodes MM, Heiny ME, Fuh B, Fixler JM, Gordon MO, DeBaun MR. Silent cerebral infarction, income, and grade retention among students with sickle cell anemia. Am J Hematol. 2014 Oct;89(10):E188-92. doi: 10.1002/ajh.23805. Epub 2014 Aug 4. PMID 25042018
- [Background] Yarboi J, Compas BE, Brody GH, White D, Rees Patterson J, Ziara K, King A. Association of social-environmental factors with cognitive function in children with sickle cell disease. Child Neuropsychol. 2017 Apr;23(3):343-360. doi: 10.1080/09297049.2015.1111318. Epub 2015 Nov 15. PMID 26568287
- [Background] Hoyt CR, Varughese TE, Erickson J, Haffner N, Luo L, L'Hotta AJ, Yeager L, King AA. Developmental delay in infants and toddlers with sickle cell disease: a systematic review. Dev Med Child Neurol. 2022 Feb;64(2):168-175. doi: 10.1111/dmcn.15048. Epub 2021 Sep 17. PMID 34535892
- [Background] Fields ME, Hoyt-Drazen C, Abel R, Rodeghier MJ, Yarboi JM, Compas BE, King AA. A pilot study of parent education intervention improves early childhood development among toddlers with sickle cell disease. Pediatr Blood Cancer. 2016 Dec;63(12):2131-2138. doi: 10.1002/pbc.26164. Epub 2016 Aug 11. PMID 27509845
- [Background] Varni JW, Panepinto JA. Cognitive functioning, patient health communication, and worry mediate pain predictive effects on health-related quality of life in youth with sickle cell disease. Pediatr Blood Cancer. 2020 Nov;67(11):e28680. doi: 10.1002/pbc.28680. Epub 2020 Aug 29. PMID 32860648
- [Background] Hardy SJ, Bills SE, Wise SM, Hardy KK. Cognitive Abilities Moderate the Effect of Disease Severity on Health-Related Quality of Life in Pediatric Sickle Cell Disease. J Pediatr Psychol. 2018 Sep 1;43(8):882-894. doi: 10.1093/jpepsy/jsy019. PMID 29659914
- [Background] Barakat LP, Patterson CA, Daniel LC, Dampier C. Quality of life among adolescents with sickle cell disease: mediation of pain by internalizing symptoms and parenting stress. Health Qual Life Outcomes. 2008 Aug 9;6:60. doi: 10.1186/1477-7525-6-60. PMID 18691422
- [Background] Sanger M, Jordan L, Pruthi S, Day M, Covert B, Merriweather B, Rodeghier M, DeBaun M, Kassim A. Cognitive deficits are associated with unemployment in adults with sickle cell anemia. J Clin Exp Neuropsychol. 2016 Aug;38(6):661-71. doi: 10.1080/13803395.2016.1149153. PMID 27167865
- [Background] Aygun B, Parker J, Freeman MB, Stephens AL, Smeltzer MP, Wu S, Hankins JS, Wang WC. Neurocognitive screening with the Brigance preschool screen-II in 3-year-old children with sickle cell disease. Pediatr Blood Cancer. 2011 Apr;56(4):620-4. doi: 10.1002/pbc.22833. Epub 2010 Nov 11. PMID 21298749
- [Background] Farber MD, Koshy M, Kinney TR. Cooperative Study of Sickle Cell Disease: Demographic and socioeconomic characteristics of patients and families with sickle cell disease. J Chronic Dis. 1985;38(6):495-505. doi: 10.1016/0021-9681(85)90033-5. PMID 4008590
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Ohene-Frempong K, Weiner SJ, Sleeper LA, Miller ST, Embury S, Moohr JW, Wethers DL, Pegelow CH, Gill FM. Cerebrovascular accidents in sickle cell disease: rates and risk factors. Blood. 1998 Jan 1;91(1):288-94. PMID 9414296
- [Background] Piel FB, Steinberg MH, Rees DC. Sickle Cell Disease. N Engl J Med. 2017 Apr 20;376(16):1561-1573. doi: 10.1056/NEJMra1510865. No abstract available. PMID 28423290
- [Background] Hassell KL. Population estimates of sickle cell disease in the U.S. Am J Prev Med. 2010 Apr;38(4 Suppl):S512-21. doi: 10.1016/j.amepre.2009.12.022. PMID 20331952